CLINICAL TRIAL: NCT06214936
Title: The VILOCITY Trial: Validating Incubators in the Lab: Optimizing Culture and Investigating blasTulation Yield: a Randomized Control Trial (RCT)
Brief Title: Validating Incubators in the Lab: Optimizing Culture and Investigating blasTulation Yield
Acronym: VILOCITY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Collaborators: CooperSurgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2206-BRG-075-CW
Record Dates: First submitted 2023-10-25; First posted 2024-01-22 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oocytes allocated to the benchtop incubator (Other): Half of the mature oocytes and subsequent embryos will be cultured in the benchtop incubator
  Interventions: Other: Benchtop Incubator
- Oocytes allocated to the box incubator (Other): Half of the mature oocytes and subsequent embryos will be cultured in the box incubator
  Interventions: Other: Box Incubator

INTERVENTIONS:
Other: Benchtop Incubator — half of the mature oocytes will be placed in the benchtop incubator and after ICSI the resulting inseminated oocytes and subsequent embryos will remain in the benchtop incubator for the remainder of embryo culture
  Arms: Oocytes allocated to the benchtop incubator
Other: Box Incubator — half of the mature oocytes will be placed in the benchtop incubator and after ICSI the resulting inseminated oocytes and subsequent embryos will remain in the box incubator for the remainder of embryo culture
  Arms: Oocytes allocated to the box incubator

SUMMARY:
The goal of this study is to determine if benchtop incubators improve the number of embryos making it to the blastocyst stage of development (about 4-6 days after fertilization) in people undergoing in vitro fertilization (IVF) treatment for their infertility.

* Test the effectiveness of the benchtop incubator.
* Determine if the number of embryos reaching the blastocyst stage of embryo development (the stage that the embryos are biopsied for PGT-A and frozen) is improved in the benchtop incubator compared to the box incubator.
* Compare embryology outcomes between the two incubator types.
* Investigate transfer and pregnancy outcomes.
* Expand the knowledge surrounding the impact of the incubator on IVF outcomes. Patients will have their mature oocytes collected at the egg retrieval procedure split into two groups and randomized to be cultured in both incubator types.

DETAILED DESCRIPTION:
The proposed study is a prospective, split cohort, randomized controlled trial which seeks to characterize blastocyst formation rates following culture in a benchtop incubator in comparison to a box incubator. Following enrollment, participants will undergo ovarian stimulation and oocyte retrieval per routine as previously consented to at the clinic. IVF stimulation protocol will be at the discretion of the participant's individual provider, per routine. Those participants that develop 4 or more mature oocytes will proceed with randomization. Intracytoplasmic Sperm Injection (ICSI) will be performed, as well as assisted hatching on day 3 and embryos will be cultured to the blastocyst stage per routine. It is important to note that there are no changes to the routine embryology care itself, the only difference within the study is that the participant's cohort of oocytes will be split into two groups and randomized to placement within each type of incubator (benchtop and conventional box incubator). The participant, physician, and the clinical team will all be blinded to the randomization of the oocytes and subsequent embryos until study completion. All embryologists making any assessments or selecting the embryo for transfer will also be blinded.

ELIGIBILITY:
Inclusion Criteria for participants:

1. Patients undergoing an IVF cycle with plan for subsequent frozen embryo transfer (FET) of a single euploid embryo
2. 4 mature oocytes prior to randomization
3. Female partners age <42 years old at start of their vaginal oocyte retrieval (VOR) cycle
4. Normal ovarian reserve:

   1. Antimullerian Hormone Level (AMH) ≥ 1.2 ng/mL
   2. Antral Follicle Count (AFC) ≥ 8
   3. Follicle Stimulating Hormone (FSH) FSH ≤ 12international units (IU)/L
5. Body Mass Index (BMI) <35
6. Patients who desire to transfer the best quality embryo for their embryo transfer. However, if a participant ends up electing to transfer based on sex preference after enrollment these outcomes will still be followed and included in the intention to treat analysis.

Exclusion Criteria for participants:

1. All patients who do not voluntarily give their written consent for participation
2. Patients with a prior failed IVF cycle - defined as no blastocysts
3. Patients with a history of more than one failed euploid embryo transfer
4. Donor oocyte cycles
5. Gestational Carriers
6. Male partner with <100,000 total motile spermatozoa per ejaculate (donor sperm is acceptable)
7. Use of surgical procedures to obtain sperm
8. Communicating hydrosalpinges without a plan for surgical correct prior to frozen embryo transfer
9. Endometrial Insufficiency, as defined by a prior cycle with maximal endometrial thickness <6mm,), or persistent endometrial fluid
10. Single gene disorders, chromosomal translocations, or any other disorders requiring a more detailed embryo genetic analysis

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Blastulation Rate per mature oocyte (M2) | approximately 1 week post oocyte retrieval procedure
  count of blastocyst stage embryos per M2 count

SECONDARY OUTCOMES:
Fertilization Rate | approximately 24 hours post oocyte retrieval procedure
  count of fertilized zygotes (2 pronuclei (2PN)) per M2 count
Blastulation Rate per 2PN | approximately 1 week post oocyte retrieval procedure
  count of blastocyst stage embryos per 2PN
Blastocyst Morphology using Modified Gardner Scale | approximately 1 week post oocyte retrieval procedure
  Morphology Grade at time of trophectoderm biopsy and vitrification. Expansion 1-6. Inner cell mass and trophectoderm graded A-D.
Ploidy rates | approximately 2 weeks post blastocyst trophectoderm biopsy
  Rates of whole chromosome negative and positive preimplantation genetic testing for aneuploidy (PGT-A) results per blastocyst
Sustained implantation rate (SIR) | 6 weeks post embryo transfer
  rate of ongoing pregnancy at 8-9 weeks gestational age when discharged to obstetrician
Live birth rate | approximately 7 months after discharge to obstetrician
  rate of live born infants
Embryologist Questionnaire | upon primary outcome completion in approximately 18 months
  assess efficiency in the lab between the two incubators and other questions from the embryologist's perspectives

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Molinaro, MD, MSCE, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States